CLINICAL TRIAL: NCT04451564
Title: Understanding and Restoring Dopaminergic Function in Fibromyalgia Patients Using a Mindfulness-based Psychological Intervention: A [18F]-DOPA Positron Emissions Tomography (PET) Study Study Protocol for the FIBRODOPA Study- a Randomized Controlled Trial
Brief Title: Understanding and Restoring Dopaminergic Function in Fibromyalgia Patients
Acronym: FIBRODOPA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Fribourg (Other)
Collaborators: University of Lausanne (Other); University of Zurich (Other); University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: FIBRODOPA TRIAL
Record Dates: First submitted 2020-06-19; First posted 2020-06-30 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Fibromyalgia
Keywords: dopamine; reward; F-DOPA; mindfulness
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MORE Mindfulness oriented recovery enhancement group (Experimental): MORE Mindfulness oriented recovery enhancement group
  Interventions: Behavioral: Mindfulness oriented recovery enhancement
- Control (No Intervention): wait-list

INTERVENTIONS:
Behavioral: Mindfulness oriented recovery enhancement — 8- week psychological program based on mindfulness techniques
  Arms: MORE Mindfulness oriented recovery enhancement group

SUMMARY:
Fibromyalgia (FM) is a very prevalent and debilitating chronic pain disorder that is difficult to treat. Mindfulness-based techniques are regarded as a very promising approach for the treatment of chronic pain and in particular FM. The Mindfulness-Oriented Recovery Enhancement (MORE) intervention, a mindfulness-based group intervention, has shown beneficial effects in opioid-treated chronic pain patients, including reduced pain severity, functional interference, and opioid dosing, by restoring neurophysiological and behavioral responses to reward. First evidence for a hypodopaminergic state and impaired reward processing in FM have been reported. However, little is known about its impact on dopamine (DA) function and in particular with regard to DA responses to monetary reward in FM. The aim of the present study protocol is to evaluate if MORE is able to restore the DA function in FM patients, in particular with regard to the DA responses to reward, and to reduce pain and mood complaints in FM.

DETAILED DESCRIPTION:
the present study is a multi-center randomized controlled trial (RCT) with 3 time points: before the intervention, after completion of the intervention and 3-months after completion of the intervention. Eighty FM patients will be randomly assigned to either the MORE intervention (N=40) or to a wait-list control group (N=40). Additionally a comparison group of healthy women (N=20) will be enrolled. The MORE intervention consists of eight 2-hour long group sessions administered weekly over a period of 8 weeks. Before and after the intervention, FM participants will undergo [18F] DOPA Positron Emission Tomography (PET) and functional magnetic resonance (MR) imaging while performing a monetary reward task. The primary outcome will be endogeneous DA changes measured with [18F] DOPA PET at baseline, after the intervention (after 8 weeks for control group), and at 3 months' follow-up. Secondary outcomes will be (1) clinical pain measures and FM symptoms using standardized clinical scales 2) functional brain changes 3) measures of negative and positive affect, stress and reward experience in daily life using the Experience Sampling method (ESM) 4) biological measures of stress including cortisol and alpha-amylase.

Design: If the findings of this study confirm the effectiveness of MORE in restoring DA function, reducing pain and improving mood symptoms, MORE can be judged to be a promising means to improve quality of life in FM patients. The findings of this trial may inform health care providers about the potential use of the MORE intervention as a possible non-pharmacological intervention for FM.

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgia syndrome
* no psychiatric disorders
* right handed
* older than 18 years,

Exclusion Criteria:

* male sex
* history of neurological disorders
* left handed
* psychiatric disorders
* current substance or tobacco abuse
* current and past substance dependence
* schizophrenia spectrum disorder
* any other form of chronic pain apart from Fibromyalgia

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Dopamine response | within the second year
  Dopamine response measured with 18F-DOPA as percent Bold signal change Range 0.001 +/-0.009 ml g -1 per min

SECONDARY OUTCOMES:
changes in pain and clinical related measures | within the second year
  measured with the brief pain inventory questionnaire (BPI, Cleeland, 1994) Range: 0-40. 0 corresponds to no interference with pain in daily life and 40 corresponds to maximal interference of pain in daily life

CONTACTS AND LOCATIONS:
Overall Officials: Chantal o Martin Sölch, PhD, Principal Investigator — University of Fribourg
Locations (1):
- University of Fribourg, Fribourg, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ledermann K, von Kanel R, Berna C, Sprott H, Burckhardt M, Jenewein J, Garland EL, Martin-Solch C. Understanding and restoring dopaminergic function in fibromyalgia patients using a mindfulness-based psychological intervention: a [18F]-DOPA PET study. Study protocol for the FIBRODOPA study-a randomized controlled trial. Trials. 2021 Dec 1;22(1):864. doi: 10.1186/s13063-021-05798-1. PMID 35078536